CLINICAL TRIAL: NCT06945965
Title: Evaluation of Different Scaffolds in Regenerative Endodontic Treatment of Immature Non-Vital Permanent Teeth and Their Release of Growth Factors: A Randomized Clinical Trial
Brief Title: Evaluation of Different Scaffolds in Regenerative Endodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Riham Karam Ahmed, Ass.Lecturer, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Regenerative Endodontic
Record Dates: First submitted 2025-04-03; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Endodontic Disease; Regenerative Endodontics
Keywords: PRF; Regeneration; Blood Clot; Scaffolds
MeSH Terms: conditions — Dental Pulp Diseases; Thrombosis | interventions — proliferation regulatory factors, human urine; Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The trial design of this study is planned to be a double-blinded design in which the participant and the statistician will be blinded, and only the operator knows which treatment the patient will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regeneration with Injectable platelet-rich fibrin (i-PRF) scaffold (Experimental): 10 ml of venous blood was drawn from the patient's arm. Then it was collected in a sterile tube without anticoagulant.
  * The collected blood was centrifuged immediately.
  * The separated plasma and platelets form a light-yellow-colored layer, which is situated at the top of the tube. This is then aspirated using a syringe with a needle and amounts to a partially active injectable form.
  Interventions: Procedure: Injectable platelet-rich fibrin (i-PRF) scaffold
- Regeneration with platelet-rich fibrin (PRF)scaffold (Experimental): 10 ml venous blood was drawn from the patient's arm
  * Then it was collected in a sterile tube without anticoagulant.
  * The collected blood was centrifuged immediately.
  * Following the centrifugation, the fibrin clot was formed in the middle of the tube between the red corpuscles at the bottom and acellular plasma at the top.
  Interventions: Procedure: platelet-rich fibrin (PRF)scaffold
- Regeneration with blood clot (BC) scaffold (Active Comparator): The file will be passed 2 mm beyond the apical end to induce bleeding inside the canal till approximately 2-3 mm below the CEJ.
  Interventions: Procedure: blood clot (BC) scaffold

INTERVENTIONS:
Procedure: Injectable platelet-rich fibrin (i-PRF) scaffold — The separated plasma and platelets form a light-yellow-colored layer, which is situated at the top of the tube. This is then aspirated using a syringe with a needle (partially active injectable form).
  Arms: Regeneration with Injectable platelet-rich fibrin (i-PRF) scaffold
Procedure: platelet-rich fibrin (PRF)scaffold — The fibrin clot was removed from the test tube with sterile tweezers, then cut into fragments, then placed incrementally in the canal space below the CEJ using hand pluggers (without prior induction of apical bleeding).
  Arms: Regeneration with platelet-rich fibrin (PRF)scaffold
Procedure: blood clot (BC) scaffold — A sterile saline-soaked cotton pellet was placed into the canal 2 mm below the orifice for 15 minutes to form a blood clot.
  Arms: Regeneration with blood clot (BC) scaffold

SUMMARY:
The aim of this study is to evaluate and compare the regenerative potentials of Injectable Platelet-Rich Fibrin (I-PRF), Platelet-Rich Fibrin (PRF), and Blood Clot (BC) as different scaffolds regarding:

Radiographic outcomes (increase of root length, increase in thickness of dentinal wall, healing of periapical lesion, and apical closure).

Clinical outcomes in the treatment of young, immature permanent teeth with necrotic pulps.

ELIGIBILITY:
Inclusion Criteria:

* Necrotic immature permanent anterior teeth.
* Teeth not indicated for post/core final restoration.
* Radiographically: The root has incomplete development with an apical opening of more than 1 mm.

Exclusion Criteria:

* Medically compromised patients with blood and immunity disorders. Family history of autoimmune disorder. Also, patients with physical or mental handicapping conditions.
* Teeth with questionable restorability of the remaining crown/root structure.
* Pathological tooth mobility.
* Radiographically: Evidence of root fracture or root resorption (external or internal).

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Root Length | 12 months
  the distance between the CEJ and the apical endpoint mesially (M) and distally (D) on the coronal plane and labially (L) and palatally (P) on the sagittal plane. it was measured by a measure length tool in millimeters.
Root dentine thickness | 12 months
  Root dentine thickness was measured as a line from the outer root canal diameter to the canal lumen in the mesial, distal, buccal, and lingual dentinal walls of the root. It was measured from the axial plane at 4 mm and 8 mm from the CEJ. It was measured by the same length-measuring tool in millimeters.
Apical foramen diameter | 12months
  It was measured as a line from the mesial and distal root ends at the coronal plane and from the labial to palatal root ends at the sagittal plane in millimeters.
Bony lesion volume | 12 months
  The volume of each slice of the lesion was calculated by multiplying the area of each cut by the distance of 0.5mm between the tomographic sections. With the sum of the volume of all the slices, the total volume of the bony lesion was obtained in cubic centimeters.

SECONDARY OUTCOMES:
Pulp sensibility | 12 months
  response to the cold with ethyl chloride and/or electrical pulp testing.

CONTACTS AND LOCATIONS:
Overall Officials: shehab M Mohamed, Phd, Study Director — British University In Egypt
Locations (1):
- British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masuki H, Okudera T, Watanebe T, Suzuki M, Nishiyama K, Okudera H, Nakata K, Uematsu K, Su CY, Kawase T. Growth factor and pro-inflammatory cytokine contents in platelet-rich plasma (PRP), plasma rich in growth factors (PRGF), advanced platelet-rich fibrin (A-PRF), and concentrated growth factors (CGF). Int J Implant Dent. 2016 Dec;2(1):19. doi: 10.1186/s40729-016-0052-4. Epub 2016 Aug 22. PMID 27747711
- [Background] El Bagdadi K, Kubesch A, Yu X, Al-Maawi S, Orlowska A, Dias A, Booms P, Dohle E, Sader R, Kirkpatrick CJ, Choukroun J, Ghanaati S. Reduction of relative centrifugal forces increases growth factor release within solid platelet-rich-fibrin (PRF)-based matrices: a proof of concept of LSCC (low speed centrifugation concept). Eur J Trauma Emerg Surg. 2019 Jun;45(3):467-479. doi: 10.1007/s00068-017-0785-7. Epub 2017 Mar 21. PMID 28324162
- [Background] Metlerska J, Fagogeni I, Nowicka A. Efficacy of Autologous Platelet Concentrates in Regenerative Endodontic Treatment: A Systematic Review of Human Studies. J Endod. 2019 Jan;45(1):20-30.e1. doi: 10.1016/j.joen.2018.09.003. Epub 2018 Nov 13. PMID 30446403
- [Background] Murray PE. Platelet-Rich Plasma and Platelet-Rich Fibrin Can Induce Apical Closure More Frequently Than Blood-Clot Revascularization for the Regeneration of Immature Permanent Teeth: A Meta-Analysis of Clinical Efficacy. Front Bioeng Biotechnol. 2018 Oct 11;6:139. doi: 10.3389/fbioe.2018.00139. eCollection 2018. PMID 30364277